CLINICAL TRIAL: NCT03098563
Title: Maximizing Analgesia to Reduce Pain Sensitivity in Chronic Knee Osteoarthritis Pain Patients
Brief Title: Maximizing Analgesia to Reduce Pain in Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00125605; R01DA042751 (NIH)
Record Dates: First submitted 2017-03-17; First posted 2017-04-04 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis
Keywords: Clinical Trial; Phase II
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Central Nervous System Stimulants; Benzodiazepines; Analgesics, Opioid; Cannabinoids; Nonprescription Drugs; Dosage Forms

STUDY DESIGN:
Intervention Model Description: This study will include 4 sessions. Participants will be randomly assigned to the order in which they receive one drug (or combination of drugs) per session at each study visit.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Within-subjects design. Two pills will be administered at each study visit. Participants and study staff will be blind to the drug(s) administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (Experimental): Blinded study medication. This is a within-subject study so all session procedures will be identical. The specific medications administered that study day will be the only change each session. Study days will last approximately 8 hours and will be conducted on an outpatient basis. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  Interventions: Drug: Blinded study medication
- Arm 2 (Experimental): Blinded study medication. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  Interventions: Drug: Blinded study medication
- Arm 3 (Experimental): Blinded study medication. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  Interventions: Drug: Blinded study medication
- Arm 4 (Experimental): Blinded study medication. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  Interventions: Drug: Blinded study medication

INTERVENTIONS:
Drug: Blinded study medication — Blinded study medication: This is a double-blind within-subject Phase II trial. Study medications will remain blinded. Participants may receive a dose of medication from one or more of the following categories: prescription stimulants, prescription benzodiazepines, prescription opioids, prescription cannabinoids, over-the-counter medications or placebo (sugar pill). All subjects will serve as their own control. Study medication administration will be randomized within each participant.
  Other Names: stimulants, benzodiazepines, opioids, cannabinoids, over the counter (OTC) medications, placebo

SUMMARY:
This research is being done to evaluate whether combining medications that are FDA approved, but have not yet been approved for combination treatment, can be effective in reducing pain.

DETAILED DESCRIPTION:
This study will evaluate whether a combination of pharmacotherapies can effectively alleviate pain. Subjects will complete two screening sessions before completing four study sessions that will occur once weekly. Participants will receive double blind doses of study medications the morning of each experimental session day and will undergo standardized pain testing, physical functioning assessment, blood draws, ratings of drug effects and cognitive testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee osteoarthritis
* Urine sample tests negative for common illicit substances of abuse (e.g., cannabis)
* Medically cleared to take study medications
* Are not pregnant or breast feeding
* Willing to comply with the study protocol.

Exclusion Criteria:

* Pain other than Knee Osteoarthritis
* Taking opioids for pain
* Prescribed and taking gabapentinoid, Tricyclic Antidepressants (TCA), venlafaxine, duloxetine, stimulants or benzodiazepines
* Presence of any clinically significant medical/psychiatric illness judged by the investigators to put subject at elevated risk for experiencing an adverse event
* Known allergy to the blinded study medications

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Campbell, Ph.D., Principal Investigator — Johns Hopkins University; Kelly E Dunn, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Experimental Session 1 is a safety session and completed first. The remaining sessions were completed in triple blinded randomized order.
Groups:
- Hydromorphone+Placebo: Within-subject double-blind, double-dummy administration of hydromorphone (oral) + placebo. Always administered during session 1. This is a within-subject study so all session procedures will be identical. The specific medications administered that study day will be the only change each session. Study days will last approximately 8 hours and will be conducted on an outpatient basis. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  This is a double-blind within-subject Phase II trial. Study medications will remain blinded. All subjects will serve as their own control. Study medication administration will be randomized within each participant.
- Placebo+Placebo: Within-subject double-blind, double-dummy administration of placebo + placebo. Order of dose randomized session days 2-4. This is a within-subject study so all session procedures will be identical. The specific medications administered that study day will be the only change each session. Study days will last approximately 8 hours and will be conducted on an outpatient basis. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  This is a double-blind within-subject Phase II trial. Study medications will remain blinded. All subjects will serve as their own control. Study medication administration will be randomized within each participant.
- Dronabinol + Placebo: Within-subject double-blind, double-dummy administration of dronabinol + placebo. Order of dose randomized session days 2-4. This is a within-subject study so all session procedures will be identical. The specific medications administered that study day will be the only change each session. Study days will last approximately 8 hours and will be conducted on an outpatient basis. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  This is a double-blind within-subject Phase II trial. Study medications will remain blinded. All subjects will serve as their own control. Study medication administration will be randomized within each participant.
- Hydromorphone + Dronabinol: Within-subject double-blind, double-dummy administration of hydromorphone + dronabinol. Order of dose randomized session days 2-4. This is a within-subject study so all session procedures will be identical. The specific medications administered that study day will be the only change each session. Study days will last approximately 8 hours and will be conducted on an outpatient basis. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  This is a double-blind within-subject Phase II trial. Study medications will remain blinded. All subjects will serve as their own control. Study medication administration will be randomized within each participant.
Period: Experimental Session 1
Arm/Group | Hydromorphone+Placebo | Placebo+Placebo | Dronabinol + Placebo | Hydromorphone + Dronabinol
Started | 58 | 0 | 0 | 0
Completed | 58 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Experimental Sessions 2-4
Arm/Group | Hydromorphone+Placebo | Placebo+Placebo | Dronabinol + Placebo | Hydromorphone + Dronabinol
Started | 0 | 58 | 0 | 0
Completed | 0 | 58 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Experimental Sessions 2-4
Arm/Group | Hydromorphone+Placebo | Placebo+Placebo | Dronabinol + Placebo | Hydromorphone + Dronabinol
Started | 0 | 0 | 58 | 0
Completed | 0 | 0 | 58 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Experimental Sessions 2-4
Arm/Group | Hydromorphone+Placebo | Placebo+Placebo | Dronabinol + Placebo | Hydromorphone + Dronabinol
Started | 0 | 0 | 0 | 58
Completed | 0 | 0 | 0 | 58
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: This is a within-subject study so all session procedures will be identical. The specific medications administered that study day will be the only change each session. Study days will last approximately 8 hours and will be conducted on an outpatient basis. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  This is a double-blind within-subject Phase II trial. Study medications will remain blinded. All subjects will serve as their own control. Study medication administration will be randomized within each participant.
Arm/Group | Overall
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.34 (6.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 31
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Largest Change From Baseline on Clinical Pain Rating
Description: The study will measure whether blinded study medications change clinical pain ratings (0-100 pain rating scale). Higher score indicates worse outcome. Biggest difference from baseline over the entire session is reported.
Time Frame: 8 hour study session
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo + Placebo: Placebo + Placebo. This is a within-subject study so all session procedures will be identical. The specific medications administered that study day will be the only change each session. Study days will last approximately 8 hours and will be conducted on an outpatient basis. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  Blinded study medication: Placebo + Placebo. This is a double-blind within-subject Phase II trial. Study medications will remain blinded. All subjects will serve as their own control. Study medication administration will be randomized within each participant.
- Hydromorphone + Placebo: Hydromorphone + Placebo. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  Blinded study medication: Hydromorphone + Placebo. This is a double-blind within-subject Phase II trial. Study medications will remain blinded. All subjects will serve as their own control. Study medication administration will be randomized within each participant.
- Dronabinol + Placebo: Dronabinol + Placebo. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  Blinded study medication: Dronabinol + Placebo. This is a double-blind within-subject Phase II trial. Study medications will remain blinded. All subjects will serve as their own control. Study medication administration will be randomized within each participant.
- Hydromorphone + Dronabinol: Hydromorphone + Dronabinol. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  Blinded study medication: Hydromorphone + Dronabinol. This is a double-blind within-subject Phase II trial. Study medications will remain blinded. All subjects will serve as their own control. Study medication administration will be randomized within each participant.
Arm/Group | Placebo + Placebo | Hydromorphone + Placebo | Dronabinol + Placebo | Hydromorphone + Dronabinol
Number analyzed (Participants) | 58 | 58 | 58 | 58
score on a scale
  Baseline | 24.19 (23.63) | 30.48 (27.39) | 28.55 (26.78) | 26.38 (25.86)
  Peak Effect | 12.76 (17.81) | 9.40 (16.27) | 12.80 (17.50) | 12.41 (16.92)
Statistical Analysis 1: Comparison: Placebo + Placebo vs Hydromorphone + Placebo vs Dronabinol + Placebo vs Hydromorphone + Dronabinol; Test type: Superiority; p = .021, ANOVA

ADVERSE EVENTS:
Time Frame: Up to 40 hours
Groups:
- Hydromorphone + Placebo: Hydromorphone + Placebo. This is a within-subject study so all session procedures will be identical. The specific medications administered that study day will be the only change each session. Study days will last approximately 8 hours and will be conducted on an outpatient basis. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  Blinded study medication: Hydromorphone + Placebo. This is a double-blind within-subject Phase II trial. Study medications will remain blinded. All subjects will serve as their own control. Study medication administration will be randomized within each participant.
- Dronabinol + Placebo: Dronabinol + Placebo. This is a within-subject study so all session procedures will be identical. The specific medications administered that study day will be the only change each session. Study days will last approximately 8 hours and will be conducted on an outpatient basis. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  Blinded study medication: Dronabinol + Placebo. This is a double-blind within-subject Phase II trial. Study medications will remain blinded. All subjects will serve as their own control. Study medication administration will be randomized within each participant.
- Hydromorphone + Dronabinol: Hydromorphone + Dronabinol. This is a within-subject study so all session procedures will be identical. The specific medications administered that study day will be the only change each session. Study days will last approximately 8 hours and will be conducted on an outpatient basis. Participants will be asked to complete standardized pain testing procedures, do brief physical functioning testing, undergo blood draws and complete questionnaires and cognitive testing at multiple points over the course of each study visit.
  Blinded study medication: Hydromorphone + Dronabinol. This is a double-blind within-subject Phase II trial. Study medications will remain blinded. All subjects will serve as their own control. Study medication administration will be randomized within each participant.
Arm/Group | Placebo + Placebo | Hydromorphone + Placebo | Dronabinol + Placebo | Hydromorphone + Dronabinol
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58 | 0/58 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58 | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 15/58 | 10/58 | 13/58 | 21/58
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Placebo (N=58) | Hydromorphone + Placebo (N=58) | Dronabinol + Placebo (N=58) | Hydromorphone + Dronabinol (N=58)
Chills (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Headache (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Hypotensive (Cardiac disorders) | 1 | 1 | 1 | 1
Abdominal Cramps (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Blurred Vision (Nervous system disorders) | 0 | 0 | 1 | 2
Clumsy (Nervous system disorders) | 1 | 1 | 1 | 1
Confusion (Nervous system disorders) | 1 | 0 | 0 | 0
Coughing (Nervous system disorders) | 1 | 0 | 0 | 0
Diaphoresis (Nervous system disorders) | 1 | 0 | 0 | 0
Difficulty Concentrating (Nervous system disorders) | 1 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 1
Drowsiness (Nervous system disorders) | 1 | 1 | 1 | 1
Dry Mouth (Nervous system disorders) | 0 | 0 | 1 | 2
Impaired (Nervous system disorders) | 0 | 1 | 1 | 0
Itchy Eyes (Nervous system disorders) | 0 | 0 | 1 | 0
Light Headed (Nervous system disorders) | 1 | 1 | 0 | 2
Numb (Nervous system disorders) | 0 | 0 | 1 | 0
Restless (Nervous system disorders) | 0 | 0 | 1 | 2
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 1
Incontenance (Renal and urinary disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT03098563/Prot_SAP_000.pdf